CLINICAL TRIAL: NCT01630941
Title: Uncemented Total Hip Implant and Subcutaneous Injections of Denosumab for Patients With Osteoarthritis of the Hip. A Randomized Double Blind Placebo Controlled Study on the Effects on Bone Evaluated With DXA, PET/CT and Biochemical Markers
Brief Title: Effects of Denosumab on Periprosthetic Bone After Total Hip Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hans Mallmin (Other)
Responsible Party: Sponsor-Investigator, Hans Mallmin, MD, PhD, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2011-001481-18
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis, Hip; Ambulation Difficulty
Keywords: Osteoarthritis of the hip; Uncemented Total Hip Arthroplasty; DXA; BMD; PET; CT; Biochemical bone markers
MeSH Terms: conditions — Osteoarthritis, Hip; Mobility Limitation | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denosumab (Active Comparator): 1 ml (60 mg) subcutaneous injection Denosumab give in the posterior part of the upper arm after surgery followed by another injection 6 months later
  Interventions: Drug: denosumab
- saline (Placebo Comparator): 1 ml subcutaneous injection 0.9% saline give in the posterior part of the upper arm after surgery followed by another injection 6 months later
  Interventions: Drug: denosumab

INTERVENTIONS:
Drug: denosumab — Two doses of 60 mg in a solution of 1 ml, given as an subcutaneous injection with a 6 month interval
  Other Names: Prolia

SUMMARY:
The primary objective is to study the effect of Denosumab on Bone Mineral Density, Standardised Uptake Value and bone metabolism in patients with total hip arthroplasty. The primary hypothesis is to demonstrate that Denosumab is superior to placebo.

DETAILED DESCRIPTION:
A clinical study with 64 patients, age 35-65 years, with unilateral osteoarthritis of the hip, randomised to two groups of patients, either receiving Denosumab or placebo

The patients will operated with an uncemented total hip arthroplasty with a Continuum acetabular cup with trabecular surface (Tantalum) and longevity Highly Cross-linked Polyethylene liner, Zimmer, Warsaw, IN, USA, and a CFP femoral stem with Titanium surface and a chrome cobalt 28 mm head, Waldemar Link, Hamburg, Germany.

Clinical outcome evaluated by Harris Hip Score and EQ-5D, Bone Mineral Density by DXA, Standardised Uptake Value of Fluoride tracer, by PET/CT and biochemical markers for bone formation and bone resorption will be analyzed together with conventional radiology for implant position and fixation.

ELIGIBILITY:
Inclusion Criteria:

1. male or female patient 35-65 years of age with an unilateral OAH requiring a THA and a healthy contralateral hip
2. body weight ≤110 kg or body mass index (BMI) ≤35 kg/m2
3. living in the Uppsala County
4. the eligible patients should have been given oral information, a written Patient Information and signed an Informed Consent

Exclusion Criteria:

1. on or previously have had bone-specific treatment, e.g. bisphosphonates, raloxifene, parathyroid hormone, strontium ranelate, during the last five years
2. patients on systemical corticosteroid for more than 3 months should not be considered
3. patients with diagnosed malignant disease during the last five years or known to have metastasis from malignant disease should be excluded
4. patients with compromised general conditions and an American Society of Anesthesiologists, ASA-score >31 should not be regarded eligible
5. patients with known drug or alcohol abuse or regarded as socially dysfunctional, as judged by the investigator, should not be considered for the study
6. pregnant women or women planning for pregnancy or fertile women (premenopausal) without contraceptives should not be accepted for the study
7. patients that have been exposed frequently and/or have had large irradiation doses, as judged by the investigator, must not be included in the study.
8. enrolled in either another investigational drug study, in another investigational device study, or in another investigational study of an approved drug within 30 days prior to Visit 1 of the current study
9. any condition or laboratory findings which in the opinion of the Investigator makes the patient unsuitable for inclusion (for example claustrophobia)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-08-07 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | 12 months
  Bone mineral density by DXA in Gruen Zone 7 and a sum of Gruen zone 1-7

SECONDARY OUTCOMES:
Bone mineral Density | 24 months
  BMD, g/cm2, adjacent to the femur implant for Gruen Zone 1-7, 3, 6, and 24 months after surgery
Standardised Uptake value | 6 months
  fluoride isotope uptake, measured as (SUV), adjacent to the femoral stem, 3 and 6 months after surgery.
Standardised Uptake value | 6 months
  fluoride isotope uptake, measured as SUV adjacent to the acetabular cup 3 and 6 months after surgery
Bone Mineral density | 24 months
  BMD adjacent to the acetabular cup during the follow up period, i.e. after 3, 6, 12 and 24 months
Bone Mineral Density | 24 months
  BMD at the lumbar spine and at the contra lateral nonoperated hip 6, 12 and 24 months after surgery
Standardised Uptake Value | 6 months
  Fluoride isotope uptake measured as SUV at the lumbar spine and at the contra lateral nonoperated hip after 3 and 6 months
Biochemical markers for bone metabolism | 24 months
  biochemical markers for bone turnover and the relation to SUV and BMD findings at the proximal femur and acetabulum during the follow up period, i.e. 3, 6, 12 and 24 months after surgery
Biochemical markers for bone metabolism in relation to Bone Mineral Density and Standardised Uptake Value | 24
  biochemical markers for bone turnover and the relation to SUV and BMD findings at anatomical sites not exposed to surgery, i.e. the lumbar spine and the contra lateral hip 3 and 6 months after surgery
Biochemical markers for bone metabolism in relation to Bone Mineral Density and Standardised Uptake Value | 24
  to evaluate the natural course of an uncemented THA on BMD, i.e. the placebo group 3, 6, 12 and 24 months after surgery, SUV i.e. the placebo group 3 and 6 months after surgery and on biochemical markers, i.e. the placebo group 3, 6, 12 and 24 months after surgery
Clinical outcome evaluation | 24 months
  to evaluate the patients Quality of Life, measured by Harris Hip score and EQ-5D questionnaires
Adverse events | 24 months
  incidence and severity of adverse events (AEs) during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Hans Mallmin, MD, PhD, Principal Investigator — Uppsala University; Nils Hailer, MD, PhD, Study Chair — Uppsala University
Locations (1):
- Department of Orthopedics, Uppsala, Sweden

REFERENCES:
- [Derived] Kultima K, Ashtiani SH, Erngren I, Khoonsari PE, Carlsson H, Herman S, Freyhult E, Mallmin H, Hailer NP. Uncemented hip arthroplasty and denosumab: increased postoperative dipeptide concentrations and identification of potential new bone turnover biomarkers. JBMR Plus. 2025 May 19;9(7):ziaf091. doi: 10.1093/jbmrpl/ziaf091. eCollection 2025 Jul. PMID 40584156
- [Derived] Nystrom A, Kiritopoulos D, Ullmark G, Sorensen J, Petren-Mallmin M, Milbrink J, Hailer NP, Mallmin H. Denosumab Prevents Early Periprosthetic Bone Loss After Uncemented Total Hip Arthroplasty: Results from a Randomized Placebo-Controlled Clinical Trial. J Bone Miner Res. 2020 Feb;35(2):239-247. doi: 10.1002/jbmr.3883. Epub 2019 Nov 4. PMID 31589776